CLINICAL TRIAL: NCT05178901
Title: A Phase 1 Randomized, Single Center, Double-Blind, Placebo-Controlled, Dose-Response and Open-Label or Single Blind Booster Study to Evaluate the Safety and Immunogenicity of RVSV-Nipah Virus Vaccine Candidate PHV02 in Healthy Adult Subjects
Brief Title: A Phase 1 Study to Evaluate Safety & Immunogenicity of RVSV-Nipah Virus Vaccine Candidate PHV02 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Public Health Vaccines LLC (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PHV02-C-101
Record Dates: First submitted 2021-12-06; First posted 2022-01-05 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-01

CONDITIONS: Nipah Virus Infection
Keywords: henipavirus; vesicular stomatitis vector; paramyxoviridae infection; zoonotic disease
MeSH Terms: conditions — Henipavirus Infections; Paramyxoviridae Infections; Zoonoses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind for placebo-controlled portion; open label for Booster advance subset; single blind for remaining Booster
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- PHV02 2x10^5 pfu (Experimental)
  Interventions: Biological: PHV02
- PHV02 2x10^6 pfu (Experimental)
  Interventions: Biological: PHV02
- PHV02 2x10^7 pfu (Experimental)
  Interventions: Biological: PHV02
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- PHV02 5x10^8 pfu (Boost) (Experimental)
  Interventions: Biological: PHV02
- PHV02 5x10^8 pfu (Prime) (Experimental)
  Interventions: Biological: PHV02

INTERVENTIONS:
Biological: PHV02 — live, recombinant virus consisting of vesicular stomatitis virus (VSV; Indiana) with the gene for the Zaire ebolavirus glycoprotein (GP) (EBOV GP) replacing the gene for the VSV GP; in addition, the Nipah virus (NiV) G protein is also inserted and expressed. The vaccine is administered as a single intramuscular injection
  Arms: PHV02 2x10^5 pfu; PHV02 2x10^6 pfu; PHV02 2x10^7 pfu; PHV02 5x10^8 pfu (Boost); PHV02 5x10^8 pfu (Prime)
Other: Placebo — Lactated Ringer's Solution. The placebo will be administered as a single intramuscular injection
  Arms: Placebo

SUMMARY:
A Phase 1 Study to Evaluate the Safety and Immunogenicity of rVSV-Nipah Virus Vaccine Candidate PHV02 in Healthy Adult Subjects

DETAILED DESCRIPTION:
A Phase 1 Randomized, Single Center, Double-Blind, Placebo-Controlled, Dose-Response Study to Evaluate the Safety and Immunogenicity of rVSV-Nipah Virus Vaccine Candidate PHV02 in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

* For Booster cohort only: received PHV02 (or placebo)
* Healthy, adult, male or non-pregnant, non-lactating females
* Given written informed consent
* No clinically significant health problems
* Agree to avoid conception through Day 29
* Agree to minimize blood and body fluid exposures to others after vaccination through Day 29
* Agree to avoid exposure to immunocompromised persons after vaccination through Day 29
* Agree to avoid employment in industry involved with livestock after vaccination through Day 29

Exclusion Criteria:

* Signs or symptoms of acute COVID-19 within 1 week before vaccination.
* Prior infection with Nipah virus or suspected Henipavirus
* Healthcare worker with direct physical contact with patients
* Childcare worker in direct contact with children 5 years old or younger
* Household contact who is immunodeficient, or on immunosuppressive medication
* Hands-on food preparation job
* Primary care or treatment of cattle, horses, llamas or swine
* Hepatitis B, hepatitis C, HIV-1, HIV-2, diabetes, atopic dermatitis (eczema), chronic inflammatory disease, autoimmune or autoinflammatory disorder, malignancy, chronic or active neurologic disorder, ;
* History of severe reactions to any vaccine or history of severe allergies
* Receipt of another investigational vaccine within 30 days or a licensed vaccine within 14 days (live vaccine within 30 days)
* Known allergy to components of PHV02
* Injection sites obscured by tattoos or physical condition
* Significant psychiatric or medical condition or laboratory abnormality on screening
* History of Guillain Barre Syndrome or any chronic or acute neurological disorder
* Alcohol or illicit drug abuse within past 5 years
* Pregnant or lactating female
* Administration of blood or IgG within 120 days preceding study
* History of blood donation within 60 days of study
* Unwilling to undergo diagnostic evaluation of rash (skin biopsy, if indicated) or joint symptoms (athrocentesis if indicated by joint effusion), in both cases if acceptable to subject
* History of chronic autoimmune/autoinflammatory disease
* Elective surgery planned during the study period
* Subjects who have not adhered to and do not agree to adhere to local and institutional guidelines for COVID-19 prevention or testing
* Any subject from the Pioneer/Full cohort who experienced a hypersensitivity reaction to study vaccine or a single clinically significant Grade 3 adverse event or serious adverse event, unless deemed unrelated to vaccination, will be followed for safety and immunogenicity, but will not be eligible to enter the Booster Cohort

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by the Toxicity Grading Scale | 42 days after vaccination
  for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials
Number of participants with Nipah-specific antibody and neutralizing antibody responses as assessed by ELISA | 29 days after vaccination
  for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Monath, MD, FASTMH, Study Director — Crozet BioPharma; Carlos Fierro, MD, Principal Investigator — Johnson County Clinical Trials
Locations (1):
- Johnson County Clin-Trials(JCCT), Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No